CLINICAL TRIAL: NCT06405321
Title: Conversion or Neoadjuvant Therapy in Hepatocellular Carcinoma: A Multicenter Retrospective Study in Guangxi, China (GUIDANCE)
Brief Title: Conversion or Neoadjuvant Therapy in Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Principal Investigator, Guangxi Medical University
Other Study IDs: GUIDANCE
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: conversion therapy; neoadjuvant therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Conversion or Neoadjuvant Therapy: Patients with hepatocellular carcinoma received conversion or neoadjuvant therapy.
  Interventions: Drug: Conversion or neoadjuvant therapy.

INTERVENTIONS:
Drug: Conversion or neoadjuvant therapy. — Patients with hepatocellular carcinoma received conversion or neoadjuvant therapy.

SUMMARY:
This multicenter retrospective study which included patients with hepatocellular carcinoma (HCC) who received conversion or neoadjuvant therapy to explore the best treatment options and the best benefit group.

DETAILED DESCRIPTION:
More than 50% patients with initial hepatocellular carcinoma (HCC) are diagnosed as intermediate or advanced stage diease. Transarterial chemoembolization and systemic therapy are main treatments for these patients. With the rise of targeted drugs and immunotherapy, more and more patients with advanced HCC have access to curative treatment, thereby extending their overall survival time. In clinical practice, there are many combinations used to treat these patients. However, the safety and efficacy of conversion or neoadjuvant therapy in HCC patients remains controversial.

The aim of this project is to establish a multicentre database from Guangxi province, China, to include as many HCC patients receiving conversion or neoadjuvant therapy as possible. HCC patients who received conversion or neoadjuvant therapy as initial treatment, including hepatic artery infusion chemotherapy (HAIC), transcatheter arterial chemoembolization (TACE), tyrosine kinase inhibitors (TKIs), immune checkpoint inhibitors (ICIs), or radiotherapy were retrospectively enrolled. The purpose of this project is to explore the best beneficiaries of conversion or neoadjuvant therapy, the best treatment strategy, and the follow-up treatment options after successful conversion therapy. The ultimate objective is to provide evidence for the necessity and feasibility of conversion or neoadjuvant therapy for patients with HCC.

The data for this study were derived from the database of the regional registry platform entitled "Guangxi Liver Cancer Clinical Study Alliance (GUIDANCE)" sponsored by the Guangxi Anticancer Association Liver Cancer Committee. All of the included patients were not previously reported and were not enrolled in those industry-sponsored clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or clinically confirmed diagnosis of HCC.
* Patients who received conversion or neoadjuvant therapy as initial treatment, including hepatic artery infusion chemotherapy (HAIC), transcatheter arterial chemoembolization (TACE), tyrosine kinase inhibitors (TKIs), immune checkpoint inhibitors (ICIs), or radiotherapy.
* Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 or 1.
* With Child-Pugh 5~7 scores.

Exclusion Criteria:

* Concurrent with other malignancies within 5 years.
* Incomplete medical data.
* Follow-up time less than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma who received conversion or neoadjuvant therapy as initial treatment would be included.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  1 year overall survival

SECONDARY OUTCOMES:
progression-free survival | 1 year
  1 year progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Hong Zhong, Ph.D, Principal Investigator — Guangxi Medical University Cancer Hospital
Locations (1):
- Jian-Hong Zhong, Nanning, China, China

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available on request from the corresponding author, Jian-Hong Zhong, upon reasonable request.
Supporting Information: Study Protocol, CSR
Time Frame: After papers were published.

REFERENCES:
- [Result] Yang DL, Yan YH, Lai YC, Wu MS, Dong XF, Chen YZ, Li WF, Yang FQ, Yang YY, Zhong TM, Wang GD, Pang QQ, Chen K, Peng N, Nong JL, Su Z, Yu YQ, Ye L, Zeng FJ, Liu SP, Wang XY, Yao HB, Qin C, Zhang YY, Liu J, Li MJ, Liang YR, Wu PS, Li FX, Mao XS, Chen SC, Ou JJ, Luo M, Lu SC, Li ZC, Huang S, Su JY, Chen H, Zhang YG, Liang XM, Ma YL, Ma L, Zhong JH; GUIDANCE investigators. Prognostic value of radiological and pathological complete response following immune-based conversion therapy in patients with unresectable hepatocellular carcinoma (GUIDANCE004). JHEP Rep. 2025 Sep 8;7(11):101587. doi: 10.1016/j.jhepr.2025.101587. eCollection 2025 Nov. PMID 41143241
- [Result] Yang DL, Peng N, Nong JL, Chen K, Su Z, Yu YQ, Ye L, Zeng FJ, Liu SP, Yan YH, Wang XY, Yao HB, Yang FQ, Li WF, Qin C, Wu MS, Yang YY, Dong XF, Li MJ, Liu J, Liang YR, Wu PS, Zhong TM, Lai YC, Chen YZ, Pang QQ, Wang GD, Li FX, Mao XS, Chen SC, Ou JJ, Huo RR, Liang XM, Xiang BD, Ma L, Zhong JH; GUIDANCE Investigators. Survival Benefit of Hepatectomy after Complete or Partial Response to Conversion Therapy in Unresectable Hepatocellular Carcinoma (GUIDANCE003): A Multicenter Study. Liver Cancer. 2025 Apr 23;14(6):687-703. doi: 10.1159/000546052. eCollection 2025 Dec. PMID 40496213
- [Result] Yang DL, Ye L, Zeng FJ, Liu J, Yao HB, Nong JL, Liu SP, Peng N, Li WF, Wu PS, Qin C, Su Z, Ou JJ, Dong XF, Yan YH, Zhong TM, Mao XS, Wu MS, Chen YZ, Wang GD, Li MJ, Wang XY, Yang FQ, Liang YR, Chen SC, Yang YY, Chen K, Li FX, Lai YC, Pang QQ, Liang XM, You XM, Xiang BD, Yu YQ, Ma L, Zhong JH; GUIDANCE investigators. Multicenter, retrospective GUIDANCE001 study comparing transarterial chemoembolization with or without tyrosine kinase and immune checkpoint inhibitors as conversion therapy to treat unresectable hepatocellular carcinoma: Survival benefit in intermediate or advanced, but not early, stages. Hepatology. 2025 Aug 1;82(2):357-369. doi: 10.1097/HEP.0000000000001229. Epub 2025 Jan 15. PMID 39908184